CLINICAL TRIAL: NCT02233088
Title: A Pilot Study of a Lifestyle Intervention on the Metabolic Syndrome
Brief Title: A Pilot Study of a Lifestyle Intervention on the Metabolic Syndrome (3ELM Study)
Acronym: 3ELM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11111701-CA01; R56HL118343-01A1 (NIH)
Record Dates: First submitted 2014-08-29; First posted 2014-09-08 (Estimated); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Metabolic Syndrome
Keywords: Prediabetic State; Hypertension; Enlarged Waist Elevated Triglycerides; HDL Cholesterol, Low Serum
MeSH Terms: conditions — Metabolic Syndrome; Prediabetic State; Hypertension; Hypertriglyceridemic Waist; Hypoalphalipoproteinemias

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ELM Group (Experimental): A 6-month group lifestyle intervention, consisting of 12 weekly and 6 bi-weekly 2-hour sessions. The sessions consist of 30-min physical activity, 30-min meal demonstration, and 60-min group behavioral intervention, with a focus on experiential learning in naturalistic setting. Sessions are facilitated by dietitian/personal trainer and behavioral specialist.
  Interventions: Behavioral: ELM Group
- ELM Classes (Other): A 6-month health education, consisting of 12 weekly and 6 bi-weekly 30-45 min sessions. The sessions consist of didactic classes, with a focus on health education curriculum. Sessions are facilitated by a health educator and medical providers.
  Interventions: Other: ELM Classes
- ELM Individual (Active Comparator): A 6-month intervention, that consists of educational manuals on physical activity, diet and stress reduction and recommended 3 medical visits every 3 months for medical counseling and feedback using 5A (Ask, Advise, Assess, Assist, and Arrange) framework . These Metabolic syndrome care materials and provider documentation will be embedded in electronic medical record system, and will be accessible to medical providers by usual means. This enhanced usual care by participant's usual health care provider focuses on metabolic syndrome and lifestyle modifications to reduce the risk of chronic disease.
  Interventions: Other: ELM Individual

INTERVENTIONS:
Behavioral: ELM Group — ELM participants are trained to portion their meals according to the "Perfect Plate" method, a modified version of the USDA's ChooseMyPlate.gov. The stress management focuses on mindful living, cognitive restructuring; the enhancement of positive emotions. The physical activity component focuses on reduction of sedentary activity (by increasing daily step counts) and moderate-to-vigorous physical activity.
  Other Names: ELM Lifestyle Intervention
  Arms: ELM Group
Other: ELM Classes — ELM classes will be administered through Rush Generations program and focus on health education.
  Other Names: Health Education
  Arms: ELM Classes
Other: ELM Individual — ELM Individual arm participants will receive education materials on metabolic syndrome and diet, exercise, stress reduction recommendations. The participants will be recommended to follow these guidelines and discuss/seek support from their health care provider (visits at baseline, 3 and 6 months will be recommended.
  Arms: ELM Individual

SUMMARY:
Approximately 24% of the US adult population meet criteria for metabolic syndrome (MetS), diagnosed by a combination of abdominal obesity, elevated blood pressure, high triglyceride and low HDL-cholesterol level, and pre-diabetes. MetS quintuples the risk of diabetes, and doubles the risk of cardiovascular disease (CVD), particularly heart failure. Lifestyle modification is the initial step of treatment, but few studies have demonstrated early and sustained efficacy in remission of MetS. Our preliminary studies of a lifestyle change program for patients with MetS included a 1-year of development of an intervention by an interdisciplinary team of experts in medicine and the behavioral sciences. The investigators then tested the efficacy of the intervention in a treatment-only, proof-of-concept study. The investigators achieved our goal of 50% MetS remission after 2 years, in a sample of 26 patients. This study is the second step of a research program testing an innovative bio-behavioral intervention aimed at remitting MetS through lifestyle intervention, by focusing on eating patterns, daily activity, and stress management. The overarching objective of this research program is to determine the efficacy of the ELM lifestyle intervention to achieve remission of MetS. This purpose of the current study is to prepare for a large, randomized, clinical trial by conducting a smaller clinical trial that examines the acceptability of the ELM intervention (ELM Group) as compared to two other intervention arms (ELM Classes, ELM Individual).

DETAILED DESCRIPTION:
The 3ELM ("Eat, Love, Move") study recruits 48 patients with MetS, and provides a 6-month intervention that aims to remit MetS by promoting the long-term adoption of healthier behaviors (diet, physical activity, stress reduction). Participants in 3ELM are randomly assigned to one of the study arms ("ELM Groups", "ELM Classes", "ELM Individual"); all of which receive some type of intervention in either group, class, or individual formats. The primary aim of this project is to pilot test the acceptability of each of the study arms and the outcome measures.

The study also includes outcome assessments at 3 time points: at the start of the study, and at 3, and 6 months post baseline. All study participants will receive medical care (including metabolic syndrome care) from their regular medical doctors. Study staff will track participants' use of health care and wellness services during the study after obtaining participant permission to collect this data.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18-72 years (children and the elderly need age-specific lifestyle tailoring).
* Able to walk 2 blocks (the patients should be able to engage in moderate intensity exercise).
* Have preference for making lifestyle changes to treat MetS.
* Able to participate in a lifestyle intervention for 6 months.
* Meet at least 3 Metabolic syndrome criteria: abdominal obesity (waist girth >102♂/88♀ cm), high blood pressure (≥130/85 mm Hg or treatment), triglyceridemia (≥150 mg/dL or fibrate therapy), low HDL-cholesterol (<40♂/50♀ mg/dL or niacin therapy) or fasting glucose ≥100 mg/dL (or pre-diabetes).

Exclusion Criteria:

* Substance abuse within the past 12 months: alcohol use, current daily smokers (self-report); and illicit drug use.
* Weight loss, exceeding 10% of initial weight, in the past 6 months or current use of medications for weight loss, bowel resection surgery, bariatric surgery, eating disorder.
* Other medical or behavioral limitations judged to interfere with study participation or the ability to follow study procedures (eg, scheduled surgery, travel plans or scheduling difficulties that do not permit full participation), limited English language, cognitive impairment, pregnancy, or psychiatric comorbidities (such as severe major depression, or psychotic disorders).

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-09-20 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
metabolic syndrome remission, defined as <3 of the 5 standard diagnostic criteria. | 6-month change
  metabolic syndrome remission will be assessed by measurement of waist girth, blood pressure, fasting serum lipid and glucose levels, and the number of medications to treat blood pressure.

SECONDARY OUTCOMES:
Nutrition intake | Baseline, and 6 months
  Healthy Eating Index (HEI-2010) will be computed using data from 24-h dietary recalls, conducted on nonconsecutive days, including one weekend day, using the Nutrition Data System for Research (NDSR).128 The HEI-2010 is a quantifiable method of assessing the adherence to Dietary Guidelines for Americans.
Accelerometry | At baseline and 6 months
  Accelerometry (Actigraph) is the gold standard objective method for daily activity data collection. Standard methods for equipment programming and data reduction, supplemented by activity and sleep log will be used to calculate minutes/week of moderate/vigorous activity, sedentary activity, sleep, and accelerometer step counts.
International Physical Activity Questionnaire (IPAQ) | At baseline and 6 months
  Measures engagement in physical activity
Perceived Stress Scale | At baseline, 3, and 6 months
  a 10-item questionnaire that measures stress
Weight | At baseline, 3, and 6 months
  Weight will be measured using stationary scale per standardized protocol.
A1c | At baseline and 6 months
  A plasma sample will be collected to measure HbA1c.
Credibility and expectancies questionnaire (CEQ) | At baseline, 3, and 6 months
  A 4-item questionnaire measures participants acceptability ratings - specifically whether they think the treatments are credible and if they think they will help them with their health goals.
Vitality Index | At baseline, 3, and 6 months
  will be tracked using a 4 item subscale of Medical Outcomes Study (MOS) 36-Item Short Form Health survey that measures perceived energy and fatigue within the last 30 days.
Continuous metabolic syndrome score | At baseline, 3, and 6 months
  calculated as a sum of z-scores of the individual 5 MetS components using reported methodology from other clinical trials. This MetS research tool has methodological advantage accounting for severity of MetS.

OTHER OUTCOMES:
Medication questionnaire | At baseline, 3, and 6 months
  The list of medications with dose and frequency of administration will be collected using a standardized questionnaire.
Brief COPE | At baseline, and 6 months
  measures coping of stressors
Daily Hassles Questionnaire | At baseline, 3, and 6 months
  measures primary and secondary appraisal of stressors.
Three Factor Eating Questionnaire (TFEQ) | At baseline, and 6 months
  Measures disordered eating patterns.
Patient Health Questionnaire (PHQ-9) | At baseline, 3, and 6 months
  Measures depressive symptoms
Treatment Self-Regulation Questionnaire (TSRQ for eating and physical activity) | At baseline, 3, and 6 months
  Measures self-regulation abilities for eating and physical activity
Work Productivity and Activity Impairment Questionnaire | At baseline, 3, and 6 months
  measures lost productivity in the form of absenteeism and presenteeism.
Use of wellness, health, and preventive services | At baseline, 3, and 6 months
  Wil be used for cost analysis.
Perceived environment (food and exercise) | At baseline
  measures the built and food environment
Global health scale | At baseline, 3, and 6 months
  Self-assessment of overall health.
General Questionnaire | At baseline, updated at 3, and 6 months
  Measures basic sociodemographic characteristics.
Weight history and experiences with wellness/weight management programs | At baseline, and updated at 3 and 6 months
  Captures weight fluctuations and participation in commercial or health care based wellness or weight loss programs
Treatment modality preferences and willingness | At baseline and 6 months
  Captures participant preferences for lifestyle, medication, and surgical treatment modalities.
Beliefs about medications | At baseline
  Captures participant's beliefs about the usefulness and safety of medications.
Time horizon | At baseline and 6 months
  Assesses executive function
Patient Reported Outcomes Measurement Information System (PROMIS) Cognition questionnaire | At baseline and 6 months
  measures cognitive/executive function.
Perceived lifestyle change for physical activity and diet | At 3 and 6 months
  Captures participant's self-assessment of effort-related to lifestyle changes.

CONTACTS AND LOCATIONS:
Overall Officials: Rasa Kazlauskaite, MD, Principal Investigator — Rush University Medical Center; Lisa Walt, PhD, Study Director — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: What Is Metabolic Syndrome? — https://www.nhlbi.nih.gov/health/health-topics/topics/ms
- See also: What Causes Metabolic Syndrome? — https://www.nhlbi.nih.gov/health-topics/metabolic-syndrome
- See also: Who Is at Risk for Metabolic Syndrome? — https://www.nhlbi.nih.gov/health-topics/metabolic-syndrome
- See also: What Are the Signs and Symptoms of Metabolic Syndrome? — https://www.nhlbi.nih.gov/health-topics/metabolic-syndrome
- See also: How Is Metabolic Syndrome Diagnosed? — https://www.nhlbi.nih.gov/health-topics/metabolic-syndrome
- See also: How Is Metabolic Syndrome Treated? — https://www.nhlbi.nih.gov/health-topics/metabolic-syndrome
- See also: Living With Metabolic Syndrome — https://www.nhlbi.nih.gov/health-topics/metabolic-syndrome
- Available data/document: Clinical Study Report: PMC6589338 — https://www.ncbi.nlm.nih.gov/pubmed/30234352 — A manuscript summarizing the development of the intervention.
- Available data/document: Informed Consent Form: 11111701-IRB01 — https://rrp.rush.edu/researchportal/sd/ResourceAdministration/Project/PrintSmartForms?Project=com.webridge.entity.Entity%5BOID%5B4B88F935265BF94D8A92A0BD5A70A202%5D%5D&rootEntity=com.webridge.entity.Entity%5BOID%5B4B88F935265BF94D8A92A0BD5A70A202%5D%5D&PrintBySection=False&PrintHeaderView=True&PrintHeaderInfo=True&PrintPageBreak=True&PrintLogo=True&showHiddenData=False&showCDTFormsAtEnd=True — The informed consent is available through RuMC IRB portal.

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2014-08-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT02233088/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2013-08-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT02233088/SAP_001.pdf